CLINICAL TRIAL: NCT04739735
Title: Effectiveness of Computer - Controlled Intraligamentary Local Anaesthesia In Extraction of Mandibular Primary Molars: Randomised Controlled Clinical Trial
Brief Title: Computer - Controlled Intraligamentary Local Anaesthesia In Extraction of Primary Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Rodaina Helmy, Instructor, Pediatric Dentistry and Dental Public Health Department,Faculty of Dentistry, Alexandria University, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00010556 - 0008839
Record Dates: First submitted 2021-01-26; First posted 2021-02-05 (Actual); Results first posted 2022-01-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-11

CONDITIONS: Local Anaesthetic Drug Adverse Reaction
Keywords: Computer - controlled; Intraligamentary; Local anesthesia; Nerve block; Articaine; Pain; Extraction
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: The study will be a two-arm randomized controlled clinical trial. It will be setup and reported according to the CONSORT guidelines.
  Participants will be randomly and equally allocated to one of the two arms (Figure 1).
  * Group I: (experimental group n = 25) assigned to CC-ILA.
  * Group II: (control group n = 25) assigned to conventional injection by IANB.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The researcher (operator) who will perform all the injections and extractions as well as record heart rate measurements cannot be blinded to the type of intervention; a second impartial observer (evaluator) will record the Sensory, Eye, Motor (SEM) scale independently. The statistician will be blinded to the treatment groups. Since the participants will also be blinded, therefore, the study will be triple-blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computer Controlled -Intraligamentary Anaesthesia (CC-ILA) (Experimental): CC-ILA will be administered using the Wand-STA system according to the manufacturer instructions, It works with standardised 1.8 mL local anaesthetic carpules. The distalingual and mesiolingual line angles are the most effective for multi-rooted mandibular teeth.
  Articaine hydrochloride 4% with 1:100,000 epinephrine will be injected for each root as shown on a special indicator.The dentist will wait 5 seconds before needle withdrawal. Same steps will be repeated at the mesiolingual line angle.
  Interventions: Procedure: Dental Local Anaesthesia
- Conventional Injection of Inferior Alveolar Nerve Block (Active Comparator): * In the control group, a standard technique for the Inferior Alveolar Nerve Block (IANB) will be used supplemented with long buccal infiltration for the buccal gingiva.
  * A 27-gauge disposable dental needle will be used to inject Articaine hydrochloride 4% with 1:100,000 epinephrine. The needle will be directed between the two primary molars on the opposite side of the arch, entering the tissues at the level of the occlusal plane or slightly lower until bony resistance is met.
  Approximately 1.0 mL of LA will be delivered near the inferior alveolar nerve. Two-thirds the needle length should be inserted. The needle is withdrawn, then 0.5 ml as a long buccal infiltration distal to the second primary molar is administered.
  Interventions: Procedure: Dental Local Anaesthesia

INTERVENTIONS:
Procedure: Dental Local Anaesthesia — lower primary molar teeth indicated for extraction will be given a local anaesthetic injection according to the random allocation to one of the two arms mentioned previously

SUMMARY:
Background: Exodontia poses a psychological threat for children, increasing the need for profound local anesthesia to assure painless extraction and maintain child cooperation on the dental chair. Computer-controlled Intraligamentary anesthesia (CC-ILA) affects only the tooth to be treated with minimal pressure, eliminating the side effects of other conventional techniques.

Purpose of the study: To evaluate the effectiveness of CC-ILA injection in eliminating pain during extraction of mandibular primary molars compared to inferior alveolar nerve block (IANB) technique. The null hypothesis is there will be no difference in the pain experience with the use of CC-ILA compared to the IANB in pediatric patients.

Method: The study will be a double-blind randomized controlled clinical trial, parallel design. A total of 50 healthy children aged 5-7 years, will be selected from Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Alexandria University, Egypt. Children will be selected with scores 3 or 4 Frankl behavioral rating scale. Each child selected will have at least one mandibular primary molar that is indicated for extraction. Written informed consent will be obtained from guardian. Participants will be randomly allocated into two groups according to the technique of anesthesia that will be used. Group I (test group) will receive CC-ILA, while group II (control group) will receive IANB. Heart rate will be used as vital parameter of pain, and will be recorded at base line, during injection and during extraction procedure. Pain reaction will be assessed objectively by two investigators using Sensory, Eye, Motor (SEM) scale, while subjectively the pain will be evaluated by asking the child to express his experience using a modified face scale from the Maunuksela scale.

DETAILED DESCRIPTION:
AIM OF THE STUDY

Primary aim:

• To evaluate the effectiveness of computer - controlled Intraligamentary Anaesthesia in eliminating pain during extraction of primary mandibular molars compared to Inferior Alveolar Nerve Block.

Secondary aims:

* To assess and compare the pain experience during Local Anaesthesia injection of mandibular primary molars between computer - controlled Intraligamentary Anaesthesia and conventional Inferior Alveolar Nerve Block.
* To assess and compare the pain experience during extraction of mandibular primary molars when using the two different anaesthesia techniques.
* To record the occurrence of any adverse events.

PLAN OF THE STUDY

Study design

The study will be a two-arm randomized controlled clinical trial. It will be setup and reported according to the CONSORT guidelines. The PICOT question will be: do pediatric patients aged from 5-7 years (Population; P) assigned to receive CC-ILA (Intervention; I) in comparison to inferior alveolar nerve block conventional injection (Control; C) show less pain during injection and extraction of mandibular primary molars (outcome; O) in twenty-four hours (time; T)?

Study setting and location Participants will be recruited from Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Alexandria University, Egypt.

Sample size estimation The sample size was calculated based on results obtained from previous studies of similar nature. Sample size was estimated assuming alpha error= 5% and study power= 80%. Tekin et al reported mean ± SD Sound, Eye and Motor (SEM) score = 3.93 ± 1.223 when intraligamentary anesthesia (ILA) was used, and 5.17 ± 1.891 when inferior alveolar nerve block (IANB) was used. Based on comparison of means, sample size was calculated to be 25 per group, and the total sample size required to compare the effectiveness of CC-ILA technique versus IANB during extraction of primary mandibular molars = number of groups × number per group= 2 x 25 = 50. The sample size was calculated using powerandsamplesize.com calculator.

Randomization Participants complying with the inclusion criteria will be randomly assigned using a computer-generated list of random numbers.

Allocation concealment

Each child included in the study will be given a serial number that will be used in the allocation. These numbers will be written in identical sheets of paper with the group to which each child is allocated and placed inside opaque envelopes carrying the respective names of the children. A trial independent personnel will be assigned to the role of keeping the envelopes and unfolding them only at the time of the local anesthesia injection session so that the group the child is allocated to is concealed from the outcome evaluator.

Grouping Participants will be randomly and equally allocated to one of the two arms.

* Group I: (experimental group n = 25) assigned to CC-ILA.
* Group II: (control group n = 25) assigned to conventional injection by IANB.

Blinding

The researcher (operator) who will perform all the injections and extractions as well as record heart rate measurements cannot be blinded to the type of intervention; a second impartial observer (evaluator) will record the Sensory, Eye, Motor (SEM) scale independently. The statistician will be blinded to the treatment groups. Since the participants will also be blinded, therefore, the study will be triple-blind.

Examiner reliability

* For standardization, all clinical procedures will be performed by a single operator, who will be trained and calibrated for the Wand - STA system via training sessions by an expert through the manufacturing company, as it is too complex to be applied effectively without more appropriate training. Especially, the coordination between the foot pedal handling and the syringe has shown to be difficult.
* Training on heart rate measurement using the pulse oximeter will be also planned.
* The second observer will be trained separately to assess pain using (SEM) scale by observing children undergoing dental procedures and classifying the child's behavior on videotapes. After a 7-day interval, the exercise will be repeated in order to develop an acceptable degree of examiner reliability. Intra-examiner reliability will be tested by Intraclass correlation (ICC).

Clinical Procedure

Preliminary screening visit

• Full medical and dental history will be carried out to select patients. Those patients whose parents will give their consent to participate will be examined. Proper diagnosis with thorough clinical examination, and intraoral periapical radiograph of the tooth to be extracted will be taken to ensure that the patient will match the inclusion criteria.

Patient Preparation

• The child's dental visit will be a mean of introducing dentistry and acquainting the child to the dental unit and dental instruments using 'Tell Show Do' technique. No treatment will be done to the child in order to build a strong patient-dentist relationship.

Intervention Visit

Psychological child preparation:

* The children will be told that their teeth will be put to sleep after placing some jelly and feeling a little pinch, in order to get rid of germs.
* Audible sounds will be heard while using STA in group I, so they must be informed.
* Subjects in Group II (IANB) will be told that their cheek will feel big and funny for some time.
* The procedure will be videotaped as a method of motivation to document their good behaviour.
* Patients will be positioned in supine position with the head and chest parallel to the floor and the feet slightly elevated.
* Mouth props may aid in maintaining a wide mouth opening.
* For both groups, soft tissues will be dried using (2 x 2 cm) gauze to enhance the absorption of the topical anaesthetic. Twenty percent Benzocaine topical anaesthetic gel will be used to obtund the discomfort associated with needle insertion. It will be applied at the site of needle penetration and left in contact with the soft tissues for one minute to optimise its effect.

Local Anaesthesia Administration

1. Wand-STA system:

   * In the experimental group, CC-ILA will be administered using the Wand-STA system according to the manufacturer instructions, which is also concurrent with Mittal and Chopra (2019). It works with standardised 1.8 mL local anaesthetic carpules. The distalingual and mesiolingual line angles are the most effective for multi-rooted mandibular teeth.
   * The injection is initiated by activating the STA mode when the foot control is tapped. A 30-gauge ultra-short disposable dental needle will be inserted in the PDL through the gingival sulcus at the distolingual line angle of the target tooth first, guided by constant audible tones and visual feedback. The needle should be directed approximately 30° angle to the long axis of the tooth and the bevel facing the alveolar bone. A total of 0.9 mL Articaine hydrochloride 4% with 1:100,000 epinephrine will be injected for each root as shown on a special indicator.
   * During the anaesthetic solution delivery, the visual pressure indicator will be observed as the pressure is increasing from the red into the green zone. Tissue blanching may occur, which suggests that enough LA has been delivered. Injection will be stopped by lightly tapping the foot pedal again. The dentist will wait 5 seconds before needle withdrawal. Same steps will be repeated at the mesiolingual line angle.
2. Conventional technique:

   * In the control group, a standard technique for the Inferior Alveolar Nerve Block (IANB) will be used supplemented with long buccal infiltration for the buccal gingiva. While the mouth is open as wide as possible, the index finger palpates the injection site.
   * A 27-gauge disposable dental needle will be used to inject Articaine hydrochloride 4% with 1:100,000 epinephrine. The needle will be directed between the two primary molars on the opposite side of the arch, entering the tissues at the level of the occlusal plane or slightly lower until bony resistance is met.
   * The needle is withdrawn 2mm to aspirate. Once negative aspiration is checked, the remainder of the solution is slowly deposited. The lip and/or cheek will be shaken as a method of distraction. Approximately 1.0 mL of LA will be delivered near the inferior alveolar nerve. Two-thirds the needle length should be inserted.
   * The needle is withdrawn, then 0.5 ml as a long buccal infiltration distal to the second primary molar is administered.
   * The operator will wait for 3-5 minutes before commencing dental treatment. Numbness will be tested with a dental probe on the gingiva immediately following the injection, and after each 10 seconds in case of CC-ILA and each 30 seconds in case of IANB till full numbness is declared and the time of onset of the anaesthetic effect will be noticed.
   * In both groups, extraction will be accomplished according to AAPD guidelines.Lower full crown forceps will be used to apply slow continuous palatal/lingual and buccal force allowing for the expansion of the alveolar bone to accommodate the divergent roots and reduce the risk of root fracture.
   * Care will be taken to support the mandible with the non-extraction hand.
   * If the patient suffered pain at any given time in the experimental group, the procedure will be abandoned immediately, IANB will be administered, and extraction will be carried out.
   * Post extraction instructions will be given to the patient. They will be instructed to bite on gauze with firm pressure against the surgical site for 30 minutes. They should not disturb the surgical site or rinse vigorously on the day of extraction. According to the technique used, avoid scratching, or injuring the cheek, lips, or tongue if numbness is felt. They should avoid any physical exercise on the day of extraction. Cold soft food is recommended, as well as drinks to keep the child hydrated but without using a straw.
   * Analgesics and/or antibiotics will be prescribed if required.
   * Planning for space maintenance will be considered as well. All dental injections and extractions will be administered by the same operator, who will be assisted by a trained dental assistant.

Follow up Following extraction, follow up after 24-hours will be planned via telephone calls to assess any adverse events.

ETHICAL CONSIDERATIONS The study will be conducted following the ethical principles for medical research involving human subjects in Declaration of Helsinki. Ethical approval will be obtained from the Research Ethics Committee, Faculty of Dentistry, Alexandria University before commencing the study.

The objectives, risks and benefits of the study will be explained to parents/ guardians and a signed informed consent will be obtained prior to treatment. Verbal consent will be obtained from the children before the intervention.

Parents and children will be given age-appropriate oral hygiene instructions including proper teeth brushing twice a day especially before bedtime, as well as flossing if indicated. These measures will be demonstrated on a model. A fluoridated toothpaste and a brush will be provided to each participant on the day of the treatment.

All needed treatment will be provided to the child including any restorations, space maintainers and fluoride application. Post extraction instructions will be explained well to the parents and patients to ensure good wound healing. All the possible clinical and/or adverse outcomes will be explained to the parents and they will be asked to report immediately if any of them occurs.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 5 - 7 years.
* Children free of any systemic disease or special health care need (ASA I).
* No previous bad dental experience.
* Positive or definitely positive behaviour during preoperative assessments according to the Frankl Rating Scale (score 3 or 4).
* Patients whom their mandibular primary molars are indicated for extraction:

  * Clinical signs and sympmtoms of pulp degeneration, such as swelling or sinus tracts.
  * Radiographic evidence of periapical or interradicular radiolucency.
  * Non restorable crowns.
  * Failed pulpotomies.
* Patients whose parents will give their consent to participate.

Exclusion Criteria:

* Root resorption affecting more than one third of the root length.
* Fractured roots due to trauma.
* Signs of mobility.
* Ankylosed roots.
* Active sites of pathosis in area of injection that could affect anaesthetic assessment.
* History of allergy to local anesthesia.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodaina H Helmy, Principal Investigator — Instructor, Pediatric Dentistry and Dental Public Health Department
Locations (1):
- Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
through publishing manuscripts so that other researchers could benefit from the study too.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: By August 2021
Access Criteria: it will be open access to anyone interested in research

REFERENCES:
- [Background] Maunuksela EL, Olkkola KT, Korpela R. Measurement of pain in children with self-reporting and behavioral assessment. Clin Pharmacol Ther. 1987 Aug;42(2):137-41. doi: 10.1038/clpt.1987.123. PMID 3608347
- [Background] American Academy of Pediatric Dentistry Council on Clinical Affairs. Guideline on pediatric oral surgery. Pediatr Dent. 2005-2006;27(7 Suppl):158-64. No abstract available. PMID 16541914
- [Background] Alamoudi NM, Baghlaf KK, Elashiry EA, Farsi NM, El Derwi DA, Bayoumi AM. The effectiveness of computerized anesthesia in primary mandibular molar pulpotomy: A randomized controlled trial. Quintessence Int. 2016 Mar;47(3):217-24. doi: 10.3290/j.qi.a34977. PMID 26504907
- [Background] Ran D, Peretz B. Assessing the pain reaction of children receiving periodontal ligament anesthesia using a computerized device (Wand). J Clin Pediatr Dent. 2003 Spring;27(3):247-50. PMID 12739685
- [Derived] Helmy RH, Zeitoun SI, El-Habashy LM. Computer-controlled Intraligamentary local anaesthesia in extraction of mandibular primary molars: randomised controlled clinical trial. BMC Oral Health. 2022 May 20;22(1):194. doi: 10.1186/s12903-022-02194-2. PMID 35596166
- See also: Randomisaton — http://www.sealedenvelope.com/simple-randomiser/v1/lists

RESULTS

PARTICIPANT FLOW:
Groups:
- Computer Controlled -Intraligamentary Anesthesia (CC-ILA): CC-ILA will be administered using the Wand-STA system according to the manufacturer instructions, It works with standardised 1.8 mL local anaesthetic carpules. The distalingual and mesiolingual line angles are the most effective for multi-rooted mandibular teeth.
  Articaine hydrochloride 4% with 1:100,000 epinephrine will be injected for each root as shown on a special indicator.The dentist will wait 5 seconds before needle withdrawal. Same steps will be repeated at the mesiolingual line angle.
  Dental Local Anaesthesia: lower primary molar teeth indicated for extraction will be given a local anaesthetic injection according to the random allocation to one of the two arms mentioned previously
- Conventional Injection of Inferior Alveolar Nerve Block: * In the control group, a standard technique for the Inferior Alveolar Nerve Block (IANB) will be used supplemented with long buccal infiltration for the buccal gingiva.
  * A 27-gauge disposable dental needle will be used to inject Articaine hydrochloride 4% with 1:100,000 epinephrine. The needle will be directed between the two primary molars on the opposite side of the arch, entering the tissues at the level of the occlusal plane or slightly lower until bony resistance is met.
  Approximately 1.0 mL of LA will be delivered near the inferior alveolar nerve. Two-thirds the needle length should be inserted. The needle is withdrawn, then 0.5 ml as a long buccal infiltration distal to the second primary molar is administered.
  Dental Local Anaesthesia: lower primary molar teeth indicated for extraction will be given a local anaesthetic injection according to the random allocation to one of the two arms mentioned previously
Period: Overall Study
Arm/Group | Computer Controlled -Intraligamentary Anesthesia (CC-ILA) | Conventional Injection of Inferior Alveolar Nerve Block
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Computer Controlled -Intraligamentary Aaanesthesia (CC-ILA): CC-ILA will be administered using the Wand-STA system according to the manufacturer instructions, It works with standardised 1.8 mL local anaesthetic carpules. The distalingual and mesiolingual line angles are the most effective for multi-rooted mandibular teeth.
  Articaine hydrochloride 4% with 1:100,000 epinephrine will be injected for each root as shown on a special indicator.The dentist will wait 5 seconds before needle withdrawal. Same steps will be repeated at the mesiolingual line angle.
  Dental Local Anaesthesia: lower primary molar teeth indicated for extraction will be given a local anaesthetic injection according to the random allocation to one of the two arms mentioned previously
- Total: Total of all reporting groups
Arm/Group | Computer Controlled -Intraligamentary Aaanesthesia (CC-ILA) | Conventional Injection of Inferior Alveolar Nerve Block | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Customized [Mean (Standard Deviation); unit: years] | 6.20 (0.71) | 6.00 (0.82) | 6.10 (0.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 11 | 10 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Egypt | 25 | 25 | 50
tooth location [Number; unit: teeth]
  First primary molar | 15 | 15 | 30
  Second primary molar | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Baseline Heart Rate
Description: Heart Rate will be measured using a pulse oximeter placed on child's index finger. Readings will be recorded at 2-minute intervals and the mean heart rate measurement will be calculated.
Time Frame: mean measurement when the child is seated on the dental chair until right before the injection at 2 minute intervals. time frame was approximately Minute 0 - 2
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Computer Controlled -Intraligamentary Aaanesthesia (CC-ILA) | Conventional Injection of Inferior Alveolar Nerve Block
Number analyzed (Participants) | 25 | 25
beats per minute | 99.92 (12.67) | 98.80 (15.30)

2. Primary Outcome: Heart Rate Measurement in Local Anaesthetic Administration
Description: as for outcome 1
Time Frame: starting from needle puncture till full local anaesthetic solution delivery. Time frame is approximately minute 2 - 4.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Computer Controlled -Intraligamentary Aaanesthesia (CC-ILA) | Conventional Injection of Inferior Alveolar Nerve Block
Number analyzed (Participants) | 25 | 25
beats per minute | 104.64 (12.04) | 113.48 (16.66)

3. Primary Outcome: Heart Rate Measurement in Extraction
Description: as for outcome 1
Time Frame: patient was allowed to rest for approximately 5 minutes after the injection then extraction was started. Time frame is approximately minute 9 -10
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Computer Controlled -Intraligamentary Aaanesthesia (CC-ILA) | Conventional Injection of Inferior Alveolar Nerve Block
Number analyzed (Participants) | 25 | 25
beats per minute | 107.68 (14.33) | 114.44 (19.57)

4. Primary Outcome: SEM Scale in Local Anaesthetic Administration
Description: Sound, Eye, Motor (SEM) Scale, comprises the following parameters: (1) Sound, (2) Eye, (3) Motor. For each child, the sounds, eye symptoms and body movements will be evaluated independently by a blind impartial observer using the recorded video tapes. The slightest manifestation of the sound, eyes, or motion of the patient is graded in four levels: comfort, mild, moderate, and severe discomfort, and subsequently given grades 1, 2, 3, 4, respectively. SEM score will be calculated by summing the three grades of the parameters.
Time Frame: approximately minute 2 - 4
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Computer Controlled -Intraligamentary Aaanesthesia (CC-ILA) | Conventional Injection of Inferior Alveolar Nerve Block
Number analyzed (Participants) | 25 | 25
score on a scale | 3 [3 to 4] | 9 [5 to 9]

5. Primary Outcome: SEM Scale in Extraction
Description: as for outcome 4
Time Frame: approximately minute 9 - 10
Measure: Median (Inter-Quartile Range); unit: score
Arm/Group | Computer Controlled -Intraligamentary Aaanesthesia (CC-ILA) | Conventional Injection of Inferior Alveolar Nerve Block
Number analyzed (Participants) | 25 | 25
score | 4 [3 to 8] | 7 [5 to 11]

6. Primary Outcome: Face Pain Rating Scale in Local Anaesthetic Administration
Description: A modified face scale from the Maunuksela et al scale will be used to subjectively record pain during LA injection and extraction. It consists of three schematic faces with different facial expressions for happy and sad faces representing: (A) satisfaction; (B) indifference; and (C) dissatisfaction, respectively.
Time Frame: approximately minute 2 - 4
Measure: Number; unit: participants
Arm/Group | Computer Controlled -Intraligamentary Aaanesthesia (CC-ILA) | Conventional Injection of Inferior Alveolar Nerve Block
Number analyzed (Participants) | 25 | 25
participants
  happy | 22 | 14
  indifferent | 2 | 0
  sad | 1 | 11

7. Primary Outcome: Face Pain Rating Scale in Extraction
Description: as for outcome 6
Time Frame: approximately minute 9 - 10
Measure: Number; unit: participants
Arm/Group | Computer Controlled -Intraligamentary Aaanesthesia (CC-ILA) | Conventional Injection of Inferior Alveolar Nerve Block
Number analyzed (Participants) | 25 | 25
participants
  happy | 21 | 13
  indifferent | 2 | 0
  sad | 2 | 12

8. Secondary Outcome: Assessment of Occurrence of Adverse Events
Description: Parents will be recalled after 24 hours following extraction during follow-up phone calls. Recovery parameter questions will be asked to ascertain the occurrence of lip and cheek biting, post-operative pain, or any adverse events.
Time Frame: after 24 hours
Measure: Number; unit: participants
Arm/Group | Computer Controlled -Intraligamentary Aaanesthesia (CC-ILA) | Conventional Injection of Inferior Alveolar Nerve Block
Number analyzed (Participants) | 25 | 25
participants
  Lip biting after 24 hours | 0 | 8
  Post operative pain after 24 hours | 5 | 10

ADVERSE EVENTS:
Time Frame: 4 months
Description: The present study aims to assess the children's behavioural experience while performing a routine dental procedure. There is no risk in any of the clinical interventions. Furthermore, the participants randomly selected should meet the eligibility criteria which includes a completely normal healthy patient with score ASA I in the American Society of Anesthesiologists scale.
Arm/Group | Computer Controlled -Intraligamentary Aaanesthesia (CC-ILA) | Conventional Injection of Inferior Alveolar Nerve Block
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 8/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Computer Controlled -Intraligamentary Aaanesthesia (CC-ILA) (N=25) | Conventional Injection of Inferior Alveolar Nerve Block (N=25)
lip/cheek biting (Injury, poisoning and procedural complications) | 0 (0) | 8 (8) — due to the numbness of the soft tissues caused by local anesthetic drug injection, the child could heavily bite/injure their cheeks or lower lip unconsciously, which becomes very painful after the anesthesia effect is over.

LIMITATIONS AND CAVEATS:
the children could not be blinded to the method of local anaesthesia used.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/35/NCT04739735/Prot_SAP_000.pdf